CLINICAL TRIAL: NCT04256278
Title: Does Antioxidant Administration Improve Sperm Quality in Infertile Men
Brief Title: Administration of Antioxidants to Infertile Men and Sperm Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Andrology lab Zeginiadou (Unknown); Armatura (Unknown)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Professor in Obstetrics and Gynecology and Assisted Reproduction, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHR-15
Record Dates: First submitted 2019-12-19; First posted 2020-02-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Male Infertility
Keywords: sperm; infertility; asthenospermia; oligospermia; teratozoospermia; antioxidants
MeSH Terms: conditions — Infertility, Male; Infertility; Asthenozoospermia; Oligospermia; Teratozoospermia

STUDY DESIGN:
Intervention Model Description: quadruple-blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: use of placebo, masked randomization list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Spermotrend
- Control Group (Placebo Comparator)
  Interventions: Other: Spermotrend

INTERVENTIONS:
Other: Spermotrend — oral administration of antioxidants for three months

SUMMARY:
The purpose of this randomized clinical trial is to assess the effect of oral antioxidant administration to infertile men, by evaluating semen variables, sperm DFI and levels of ROS. Oral antioxidants or placebo will be given for 3 consecutive months.

The study will recruit infertile men, who have one previous abnormal spermiogram, with at least one pathological variable (concentration, motility, morphology), according to WHO 2010 criteria. Participants will be recruited in the outpatient clinic of the Unit of Human Reproduction and of the Unit of Reproductive Endocrinology at the 1st Ob/Gyn Dept.

DETAILED DESCRIPTION:
Infertility affects up to 15% of couples trying to conceive with the male factor contributing in about 50% of cases. Oxidative stress (OS) has been found as one of the many factors causing male infertility, by inducing sperm damage. OS causes cell damage due to the raised production of reactive oxygen species (ROS), that overcome the antioxidant mechanisms of the human body. ROS are oxidizing agents that are produced as a by-product of oxygen metabolism, having at least one free electron. Due to this free electrone in their outer layer, the form very active or unstable substances. While small amounts of ROS are necessary for the proper function of sperm, increased amounts have a negative effect on sperm quality and can harm its fertility potential, thus inducing male infertility.

Spermatozoa were the first cells found to be sensitive to OS, as they lack the necessary repair cytoplasmic enzyme systems, thus being unable to repair damage. In addition, their cytoplasmic membranes are rich in polyunsaturated fatty acids (PUFAs), making them highly susceptible to oxygen-induced damage, such as lipid peroxidation (LPO). Rapid loss of intracellular adenosine triphosphate (ATP) by LPO, is responsible for axial damage, morphological damage to the sperm neck and reduced sperm motility; these events contribute to reduced sperm motility.

OS has also been associated with reduced fertilization, delayed intrauterine growth, miscarriages, birth defects (including autism) and childhood cancer. ROS found in semen come from a variety of endogenous and exogenous factors. Human sperm includes mature and immature sperm cells, leukocytes, and white blood cells. The leukocytes (mainly neutrophils and macrophages) and the immature spermatozoa are considered the major endogenous sources of ROS, whereas lifestyle, such as smoking, excessive alcohol consumption and other environmental factors such as radiation and toxins may contribute to the production of exogenous ROS.

As oxidative stress (OS) results from the imbalance of ROS overproduction and the reduced capacity of sperm antioxidant systems, many studies have aimed to improve sperm quality by administering antioxidant therapeutic regimens. In general, antioxidant therapy involves the administration of oral antioxidants, and the in vitro addition of antioxidants to culture media that are used for sample preparation in assisted reproduction techniques (ART). Many different antioxidants combinations have been studied. More and more studies have shown the beneficial effect of antioxidants on reducing sperm fragmentation and improving sperm quality. Agarwal & Sekhon's study showed a positive correlation between antioxidant therapy and various semen parameters. However, no firm conclusion regarding the beneficial effect of oral antioxidants can be made, as the majority of available studies had small sample size, used different antioxidant combinations, and the techniques that were used for the detection of ROS and DNA fragmentation index (DFI) were not standardized.

AIM OF THE STUDY The purpose of this randomized clinical trial is to assess the effect of oral antioxidant administration to infertile men, by evaluating semen variables, sperm DFI and levels of ROS.Oral antioxidants or placebo will be given for 3 consecutive months.

This study will take place at the Unit of Reproductive Endocrinology at the 1st Ob/Gyn Dept, Medical School, Aristotle University of Thessaloniki in collaboration with the private andrology diagnostic center of Mr Th. Zeginiadou.

PATIENTS The study will recruit infertile men, who have one previous abnormal spermiogram, with at least one pathological variable (concentration, motility, morphology), according to WHO 2010 criteria.

OUTCOMES

Main Outcome:

WHO Sperm analysis variable: motility.

Secondary outcomes:

WHO Sperm analysis variables: concentration, morphology. Concentration of ROS in sperm and sperm DFI.

STUDY DESIGN

Type of study:

Randomized clinical trial

The study will recruit infertile men, who have one previous abnormal spermiogram, with at least one pathological variable (concentration, motility, morphology), according to WHO 2010 criteria. Participants will be recruited in the outpatient clinic of the Unit of Human Reproduction and of the Unit of Reproductive Endocrinology at the 1st Ob/Gyn Dept. Selected participants will sign the consent form and will be asked to sample sperm at the private andrology diagnostic center of Mr Th. Zeginiadou. The sperm samples will be evaluated regarding the concentration, motility, morphology and vitality of spermatozoa, as well as the concentration of ROS, and DFI. Oral antioxidants or placebo will be given for 3 consecutive months. At the end of the 3 months period participants will be asked to re-sample their sperm in order to evaluate the same variables.

Sample size calculation Estimated sample size for two-sample means test, assuming and common standard deviation of 15 and a mean motility of 20 in the control group and 30 in the antioxidant group results in calculated sample size of 74. To allow for dropouts 80 patients will be recruited.

ELIGIBILITY:
Inclusion criteria

1. Men, 18-50 years old
2. Infertility defined as follows:

   * Failure to obtain a pregnancy after at least twelve (12) months of regular sexual intercourse without the use of contraceptives or six (6) months if the woman is> 35 years old AND
   * At least one previous abnormal spermiogram, with at least one pathological parameter (concentration, motility, morphology), according to the WHO 2010 criteria.
3. No treatment for infertility in the last three (3) months
4. Normal hormone profile (TSH, FSH, LH, total testosterone, prolactin)
5. Negative culture for mycoplasma or ureaplasma
6. Physiological scrotal ultrasound

Exclusion criteria

1. Genetic cause of infertility
2. History of cryptorchidism
3. History of orchectomy
4. History of testicular cancer
5. History of severe heart, liver or kidney disease
6. History of endocrine disease (primary or secondary hypogonadism, hyperprolactinemia, thyroid, pituitary or adrenal disease)
7. History of systemic disease or treatment in the last three (3) months
8. BMI > 30 kg/m2
9. Participation in another study and the possibility of the patient not being available for follow-up

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Sperm parameters | immediately before treatment initiation
  Sperm motility(Sperm motility was classified using a four-category scheme: A:rapid progressive, B:slow progressive, C:non-progressive, and D:immotile , %A+B, normal values >32% A+B)
Sperm parameters | immediately after the end of a 3 month treatment
  Sperm motility(Sperm motility was classified using a four-category scheme: A:rapid progressive, B:slow progressive, C:non-progressive, and D:immotile , %A+B, normal values >32% A+B)

SECONDARY OUTCOMES:
Reactive Oxygen Species (ROS) | immediately before treatment initiation
  ROS (8-hydroxy-2-deoxy-quanosine%, normal values < 3% on sperm)
Reactive Oxygen Species (ROS) | immediately after the end of a 3 month treatment
  ROS (8-hydroxy-2-deoxy-quanosine%, normal values < 3% on sperm)
DNA fragmentation Index (DFI) | immediately before treatment initiation
  DFI (%DFI: % sperm cells containing damaged DNA)
DNA fragmentation Index (DFI) | immediately after the end of a 3 month treatment
  DFI (%DFI: % sperm cells containing damaged DNA)
Sperm parameters | immediately before treatment initiation
  Sperm concentration (ml, normal values > 1.5 ml)
Sperm parameters | immediately after the end of a 3 month treatment
  Sperm concentration (ml, normal values > 1.5 ml)
Sperm parameters | immediately before treatment initiation
  Sperm morphology(Tygerberg Strict Criteria were used for the evaluation of human sperm morphology, normal form per 100 sperm, normal values >4%)
Sperm parameters | immediately after the end of a 3 month treatment
  Sperm morphology(Tygerberg Strict Criteria were used for the evaluation of human sperm morphology, normal form per 100 sperm, normal values >4%)

CONTACTS AND LOCATIONS:
Overall Officials: Stratis Kolibianakis, Professor, Principal Investigator — Aristotle University Thessaloniki
Locations (1):
- Unit of Assisted Reproduction, 1st Department of Obstetrics-Gynecology -Papageorgiou General Hospital, Thessaloniki, Greece, Thessaloniki, Central Makedonia, Greece

REFERENCES:
- [Result] Majzoub A, Agarwal A. Systematic review of antioxidant types and doses in male infertility: Benefits on semen parameters, advanced sperm function, assisted reproduction and live-birth rate. Arab J Urol. 2018 Jan 2;16(1):113-124. doi: 10.1016/j.aju.2017.11.013. eCollection 2018 Mar. PMID 29713542
- [Result] Agarwal A, Virk G, Ong C, du Plessis SS. Effect of oxidative stress on male reproduction. World J Mens Health. 2014 Apr;32(1):1-17. doi: 10.5534/wjmh.2014.32.1.1. Epub 2014 Apr 25. PMID 24872947
- [Result] Chen SJ, Allam JP, Duan YG, Haidl G. Influence of reactive oxygen species on human sperm functions and fertilizing capacity including therapeutical approaches. Arch Gynecol Obstet. 2013 Jul;288(1):191-9. doi: 10.1007/s00404-013-2801-4. Epub 2013 Mar 30. PMID 23543240
- [Result] Tremellen K. Oxidative stress and male infertility--a clinical perspective. Hum Reprod Update. 2008 May-Jun;14(3):243-58. doi: 10.1093/humupd/dmn004. Epub 2008 Feb 14. PMID 18281241
- [Result] Zini A, San Gabriel M, Baazeem A. Antioxidants and sperm DNA damage: a clinical perspective. J Assist Reprod Genet. 2009 Aug;26(8):427-32. doi: 10.1007/s10815-009-9343-5. Epub 2009 Sep 19. PMID 19768529